CLINICAL TRIAL: NCT02459912
Title: Unilateral Nerve-Sparing Cryoablation for Low-Risk, Clinically Localized, Unilateral Prostate Cancer in Potent Men: A Prospective, Phase II Trial
Brief Title: Unilateral Nerve-Sparing Cryoablation for Low-Risk, Clinically Localized, Unilateral Prostate Cancer
Acronym: POTENT-C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient recruitment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15009
Record Dates: First submitted 2015-04-29; First posted 2015-06-02 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate; Minimally; Low-Risk; Invasive; Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral Nerve-Sparing Cryoablation (Other): Unilateral Nerve-Sparing Cryoablation of the Prostate using Galil Medical Precise Cryoablation System with IceRod Needles.
  Interventions: Procedure: Unilateral Nerve-Sparing Cryoablation of the Prostate; Device: Precise Cryoablation System with IceRod Needles

INTERVENTIONS:
Procedure: Unilateral Nerve-Sparing Cryoablation of the Prostate — The side of the prostate affected by cancer will be treated with nerve-sparing cryoablation in two freeze-thaw cycles under transrectal ultrasound guidance. The unaffected side of the prostate will not be treated.
Device: Precise Cryoablation System with IceRod Needles — Galil Medical Precise Cryoablation System with IceRod Needles will be used for performing Unilateral Nerve-Sparing Cryoablation

SUMMARY:
Men with low-risk, clinically localized, unilateral prostate cancer will be treated with unilateral nerve-sparing cryoablation and evaluated for the rate of potency, cancer control and health related quality of life outcomes after treatment.

DETAILED DESCRIPTION:
This study is a clinical trial to determine and assess the change in the rate of potency in men with low-risk, localized, unilateral prostate cancer who have not received previous treatment. A total of 86 men between 40 to 69 years of age with biopsy proven, early stage localized prostate cancer will receive unilateral nerve-sparing cryoablation. The study includes a screening/pre-operative visit, a cryoablation procedure day, and 10 follow up visits over the course of 36 months. The first follow-up visit will occur within 2 weeks (±1 week) after cryoablation. Thereafter, follow-up visits will be scheduled, from the date of procedure, every 3 months (±3 weeks) for 18 months and every 6 months (±3 weeks) thereafter until the patient completes the protocol, 36 months after the cryoablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy >5 years
* Willing and able to freely sign informed consent to enroll in the study
* Willing to complete sexual function and HRQoL questionnaires
* Sexually active and potent (able to achieve an EPIC questionnaire sexual domain score greater than or equal to 75 without the use of any devices or medicines to enhance erections)
* Prostate gland volume greater than or equal to 20cc and less than or equal to 60cc
* Does not have stress urinary incontinence defined as urinary leakage requiring the use of any protective pads
* Most recent serum PSA <10 ng/mL taken at least 6 weeks after a previous biopsy and 3 months +/- 2 weeks prior to study cryoablation
* Histologically proven, clinical stage T1c-T2b prostate cancer in the proposed treated side
* Untreated contralateral side has no malignant elements demonstrated by biopsy
* Patient does not have ASAP (Atypical Small Acinar Proliferation) in the untreated side
* Patient has documented, biopsy proven unilateral disease (via a minimum of 6 biopsy cores taken on the cancerous side and a minimum of 12 negative cores on the non-cancerous side) using transrectal ultrasound (TRUS) guidance
* A 12 core biopsy using transrectal ultrasound (TRUS) guidance taken within 3 months prior to enrollment from the non-cancerous side and each core was biopsied by a site investigator
* Biopsied areas in the non-cancerous side include the following zones: L/R (left or right side) lateral base, L/R mid gland base, L/R medial base, L/R lateral middle, L/R mid gland middle, L/R medial middle, L/R lateral apex, L/R mid gland apex, L/R medial apex, L/R transitional base, L/R transitional mid, L/R anterior horn
* Prostate biopsy Gleason Score (GS) is less than or equal to 7. Gleason Score 3+4=7 [but not 4+3=7] is allowed as long as the score is based upon no more than 2 cores with cancer involvement of 50% or less.
* Does not have a biopsy GS 3+4=7 combined with clinical stage T2b
* Either a nodule was not felt (T1c) OR the palpable nodule (T2a or T2b) is on the same side as the positive biopsy

Exclusion Criteria:

* Previous treatment for prostate cancer including radiation, cryoablation, chemotherapy, surgery, high intensity focused ultrasound, and/or hormone therapy
* Previous invasive or minimally invasive treatment for benign prostatic hypertrophy (BPH) (i.e., TURP, TUMPT, WIT, TUNA)
* Inability to tolerate a transrectal ultrasound
* Active urinary tract infection
* Evidence of metastatic disease
* Irreversible bleeding diathesis or other bleeding disorders
* Anatomic penile abnormalities precluding cryoablation
* Erectile dysfunction (EPIC Questionnaire sexual domain score <60) at baseline, including the use of any erectile aid (PDE-5, etc) to increase the EPIC Questionnaire (Appendix D) sexual domain score >75, without which the patient would not qualify for the study
* Current or history within the past 6 months of alcohol and/or substance abuse which would impair participation in the study
* Major medical disorder (i.e. uncontrolled diabetes, significant hepatic, renal, or hematological disorders, recent stroke or myocardial infarction), in the opinion of the urologist, is an illness or complication which is not consistent with the protocol requirements
* Unwilling to undergo the necessary follow-up for the trial period
* Bilateral prostate cancer disease
* Significant median lobe of the prostate which would preclude an adequate cryoablation procedure (based on the discretion of the urologist)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrythmia, or psychiatric illness/social situations which would limit compliance with study requirements
* Known HIV or AIDS-related illness

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Potency Rate | 3 years
  Determine and assess the change in the rate of potency in men with unilateral prostate cancer treated with unilateral nerve-sparing cryoablation as measured by Expended Prostate Cancer Index Composite (EPIC) and International Index of Erectile Function (IIEF-15) questionnaires

SECONDARY OUTCOMES:
Cancer Control in Treated Side | 3 years
  Evaluate cancer control in the prostate side treated with unilateral nerve-sparing cryoablation by assessing the rate of tumor development
Cancer Control in Untreated Side | 3 years
  Assess the rate of tumor development in the contralateral (untreated) side of the prostate
Overall Health Related Quality of Life (EPIC) | 3 years
  Analyze the change in overall Health Related Quality of Life as measured by Expanded Prostate Cancer Index Composite (EPIC)
Overall Health Related Quality of Life (SF-12) | 3 years
  Analyze the change in overall Health Related Quality of Life as measured by the Short Form-12 (SF-12) Questionnaire
Change in Urinary Continence | 3 years
  Evaluate the change in Urinary Continence status compared to baseline as measured by the Urinary domain of the Expanded Prostate Cancer Index Composite (EPIC) questionnaire
Change in Voiding Function (IPSS) | 3 years
  Evaluate the change in voiding function compared to baseline as measured by International Prostate Symptom Score (IPSS)
Change in Voiding Function (Uroflow) | 3 years
  Evaluate the change in voiding function compared to baseline as measured by Uroflowmetry
Change in Voiding Function (PVR) | 3 years
  Evaluate the change in voiding function compared to baseline as measured by Post-Void Residual (PVR)
Change in Bowel Function | 3 years
  Evaluate the change in bowel function compared to baseline as measured by the Bowel domain of the Expanded Prostate Cancer Index Composite (EPIC) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Katz, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided